CLINICAL TRIAL: NCT02234960
Title: TOCILIZUMAB IN FIRST LINE BIOLOGIC TREATMENT OF PATIENTS WITH RHEUMATOID ARTHRITIS IN ROUTINE CLINICAL PRACTICE IN POLAND - MULTICENTER, NON-INTERVENTIONAL, PROSPECTIVE, OBSERVATIONAL STUDY (ACT-POL)
Brief Title: Local, Non-Interventional Study of RoActemra (Tocilizumab) in Poland (ACT-POL): First-Line Treatment in Routine Clinical Practice of Participants With Rheumatoid Arthritis (RA)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29444
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort of RA Participants: Participants with RA treated with tocilizumab at a dose and duration at the discretion of physician in accordance with the summary of product characteristics as per routine clinical practice were observed for a period of 6 months with the length of entire study for 24 months.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be given according to summary of product characteristics as per clinical practice.

SUMMARY:
The aim of this non-interventional, prospective, observational study is to assess the effectiveness and tolerability of RoActemra (tocilizumab) used as a first-line biologic treatment in participants with moderate to severe active RA who are inadequate responders to disease-modifying antirheumatic drugs (DMARDs), or participants who are intolerant to DMARDs, in a routine clinical practice setting in Poland. The length of the entire study will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* participants at least 18 years of age
* a diagnosis of moderate to severe RA
* treating physician has made the decision to commence tocilizumab in first line biologic treatment (population of DMARDs inadequate responders or participants who are intolerant to DMARDs) in a routine clinical practice in Poland
* informed consent

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of moderate to severe RA who are inadequate responders to DMARDs, or participants who are intolerant to DMARDs, in a routine clinical practice setting in Poland.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Remission as Assessed by Disease Activity Score 28 (DAS28 < 2.6) After 6 Months of Treatment | Month 6
Percentage of Participants with Low Disease Activity as Assessed by DAS28 (DAS28 </= 3.2) After 6 Months of Treatment | Month 6

SECONDARY OUTCOMES:
Change from Baseline in Erythrocyte Sedimentation Rate (ESR) Over Time | Baseline up to Month 6
Time to Discontinuation | Baseline up to Month 6
Percentage of Participants With Monotherapy Versus Combination Therapy with Methotrexate | Baseline up to Month 6
Percentage of Participants With Systemic Symptoms at Baseline Versus Without Systemic Symptoms at Baseline | Baseline
Percentage of Participants with Remission (DAS28 <2.6) and Low Disease Activity (DAS28 </= 3.2) After 3 Months of Treatment | Month 3
Change From Baseline in DAS28 Over Time | Baseline up to Month 6
Change From Baseline in C-Reactive Protein (CRP) Over Time | Baseline up to Month 6
Percentage of Participants With Discontinuations Due to Lack of Efficacy | Baseline up to Month 6
Percentage of Participants With Adverse Events (AEs) Or Serious AEs (SAEs) | Baseline up to Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Poland (13):
  - Bydgoszcz
  - Bytom
  - Gmina Śrem
  - Krakow
  - Lublin
  - Olsztyn
  - Poznan
  - Sieradz
  - Sopot
  - Starachowice
  - Sucha Beskidzka
  - Ustroń
  - Wroclaw